CLINICAL TRIAL: NCT06988696
Title: The Effect of Perioperative Heated Sock Application on Hypothermia and Vital Signs in Bladder Tumor Surgery:A Randomized Controlled Trial
Brief Title: The Effect of Perioperative Heated Sock Application on Hypothermia and Vital Signs in Bladder Tumor Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seval Ulubay, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Heated Sock
Record Dates: First submitted 2025-04-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Bladder Tumor
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect of Warm Sock Application on Hypothermia (Experimental): After admission to the urology ward, patients who meet the sample selection criteria will be identified one day prior to the surgical intervention. Eligible patients will be informed about the study by reading the voluntary informed consent form, which includes information about the purpose, content, and methodology of the research. Both verbal and written consent will be obtained from patients who agree to voluntarily participate in the study.
  Initially, the Descriptive Characteristics Form will be administered to the patients. One group will be given heated socks, one group will be given regular socks, and one group will not receive any intervention. The effect of these interventions on hypothermia will be examined.
  Interventions: Other: The Effect of Warm Sock Application on Hypothermia After admission to the urology ward, patients who meet the sample selection criteria will be identified one day prior to the surgical intervention.
- The Effect of Warm Sock Application on Vital Signs (Experimental): After admission to the urology ward, patients who meet the sample selection criteria will be identified one day prior to the surgical intervention. Eligible patients will be informed about the study by reading the voluntary informed consent form, which includes information about the purpose, content, and methodology of the research. Both verbal and written consent will be obtained from patients who agree to voluntarily participate in the study.
  Initially, the Descriptive Characteristics Form will be administered to the patients. One group will be given heated socks, one group will be given regular socks, and one group will not receive any intervention. The effect of these interventions on vital signs will be examined.
  Interventions: Other: The Effect of Warm Sock Application on Hypothermia After admission to the urology ward, patients who meet the sample selection criteria will be identified one day prior to the surgical intervention.

INTERVENTIONS:
Other: The Effect of Warm Sock Application on Hypothermia After admission to the urology ward, patients who meet the sample selection criteria will be identified one day prior to the surgical intervention. — The Effect of Warm Sock Application on Hypothermia After admission to the urology ward, patients who meet the sample selection criteria will be identified one day prior to the surgical intervention. Eligible patients will be informed about the study by reading the voluntary informed consent form, which includes information about the purpose, content, and methodology of the research. Both verbal and written consent will be obtained from patients who agree to voluntarily participate in the study.
  Initially, the Descriptive Characteristics Form will be administered to the patients. One group will be given heated socks, one group will be given regular socks, and one group will not receive any intervention. The effect of these interventions on hypothermia will be examined.
  Other Names: The Effect of Warm Sock Application on Vital Signs After admission to the urology ward, patients who meet the sample selection criteria will be identified one day prior to the surgical intervention.

SUMMARY:
The aim of this study is to evaluate the effect of perioperative use of heated socks on the prevention of hypothermia and its impact on vital signs in patients undergoing bladder tumor surgery. It is anticipated that the data obtained from the study will provide evidence that the use of perioperative heated socks can help prevent hypothermia and positively influence vital signs in patients undergoing bladder tumor surgery.

DETAILED DESCRIPTION:
Bladder cancer accounts for 2-3% of all malignant tumors and constitutes 6-8% of all malignancies in men and 2-3% in women. Globally, it ranks as the seventh most common cancer in men and the seventeenth in women. Bladder cancer is a significant cause of morbidity and mortality worldwide, with approximately 350,000 new cases and 150,000 deaths annually. At the time of initial diagnosis, around 75% of patients with bladder tumors are diagnosed with non-muscle-invasive bladder cancer. Of those with muscle-invasive bladder cancer, 20% are cases that have progressed from lower-stage disease. If left untreated, approximately 85% of patients with muscle-invasive bladder cancer will die from the disease . For invasive bladder tumors, the gold standard treatment is radical cystectomy. Radical cystectomy combined with pelvic lymph node dissection provides the best disease-specific survival in patients with invasive bladder tumors . Following radical cystectomy, the average 10-year disease-free survival rate is approximately 50-66%.

During the surgical process, heat loss may occur due to the evaporation of cold solutions or through perspiration. Additional factors contributing to heat loss include the patient's exposure to the operating room environment without clothing, radiation exposure, and conduction due to contact with cold materials or the stretcher. Furthermore, preoperative hypothermia, fasting, and fluid deprivation; exposure of large body surface areas during surgery; use of volatile solutions for skin preparation; evaporation of cold solutions; perspiration; major open cavity surgical interventions; administration of cold IV fluids; prolonged surgical duration and exposure to anesthesia; intraoperative blood loss; peripheral vasodilation; anesthetic drugs; absence of clothing in the operating room; radiation; contact with cold materials or the stretcher; and impaired normal thermoregulation are all factors that may contribute to hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* The duration of surgical intervention is between 2 and 4 hours,
* Ability to read, write, understand and communicate in Turkish,
* Voluntary participation in the study,
* Does not require follow-up in intensive care before or after surgery,
* Dementia, alzheimer etc. absence of disease affecting cognitive functions,
* Absence of a disease that may affect thermoregulation due to systemic effects such as chronic obstructive pulmonary disease (COPD), cancer, intracranial benign/malignant tumor, epilepsy, multiple sclerosis, Parkinson's disease, and thyroid-related diseases,
* Absence of drug use that may affect thermoregulation,
* It is not uncomfortable to wear heat socks during application.

Exclusion Criteria:

* Mental retardation and the presence of any psychiatric disorder,
* Being addicted to alcohol and drugs,
* Dementia, alzheimer etc. have a disease that affects cognitive functions,
* Having drug use that may affect thermoregulation,
* Discomfort from wearing heat socks during application,
* Having any disease that affects tissue perfusion,
* Presence of any peripheral arterial and venous disease,
* The need for intensive care before or after surgery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The Effect of Perioperative Heated Sock Application on Hypothermia and Vital Signs in Bladder Tumor Surgery:A Randomized Controlled Trial | 40 weeks
  IAs a result of the measurement in this study: Body temperature is measured tympanically. Hypothermia is generally classified based on cases where the body temperature falls below 35.0 °C. Hypothermia symptoms may vary as body temperature drops, so hypothermia is divided into three levels according to its severity.Body Temperature: Monitoring body temperature before and after surgery. Specifically, evaluating whether preoperative warm sock application helps maintain body temperature within normal ranges.
  Target Body Temperature: Assessing whether the targeted body temperature range (e.g., 36-37°C) for preventing hypothermia is achieved.

CONTACTS AND LOCATIONS:
Overall Officials: SEVAL ULUBAY, PHD, Principal Investigator — SAMSUN GAZI STATE HOSPITAL
Locations (1):
- Seval Ulubay, Samsun, Atakum/Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the approval of the board, heated socks to be used in my thesis work were obtained. Permission was granted by Samsun Gazi State Hospital, where the research would be conducted. Ethics Committee Approval was obtained from Samsun Health Sciences University Samsun Training and Research Hospital. The groups were determined through randomization over a pre-calculated sample. The pilot study is planned to begin after the randomization, and following the pilot study, necessary corrections will be made before proceeding to the data collection phase.
Supporting Information: CSR
Time Frame: August 2025-march 2026
Access Criteria: sevalulubay@gmail.com

REFERENCES:
- [Background] Lauronen SL, Kalliomaki ML, Aho AJ, Kalliovalkama J, Riikonen JM, Makinen MT, Leppikangas HM, Yli-Hankala AM. Thermal suit in preventing unintentional intraoperative hypothermia during general anaesthesia: a randomized controlled trial. Acta Anaesthesiol Scand. 2017 Oct;61(9):1133-1141. doi: 10.1111/aas.12945. Epub 2017 Jul 25. PMID 28741744